CLINICAL TRIAL: NCT02170545
Title: Computed Tomography Evaluation of Humeral Head Perfusion in Displaced Proximal Humerus Fractures in Predicting Rates of Avascular Necrosis
Brief Title: CT Imaging Evaluation of Humerus Fractures
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20000037
Record Dates: First submitted 2014-06-06; First posted 2014-06-23 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Avascular Necrosis; Humeral Fractures
Keywords: avascular necrosis; humeral head fracture; proximal arm fracture; arthroplasty
MeSH Terms: conditions — Osteonecrosis; Humeral Fractures; Shoulder Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For those patients who undergo shoulder replacement, the humeral head bone will be collected and processed for any evidence of avascular necrosis. Once processing and data collection is done, the bone will be disposed of.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multi-Part Proximal Humerus Fracture: All participants that meet the entry criteria will be included in the study cohort.
  Interventions: Other: Dual Energy Computed Tomography

INTERVENTIONS:
Other: Dual Energy Computed Tomography — A Dual Energy Computed Tomography scan will be performed on both upper arms.

SUMMARY:
Displaced, multi-part intracapsular, proximal humerus fractures represent a major challenge for patients and orthopedic surgeons. Proximal humerus fractures represent the third most common fracture after hip and distal radius fractures, and more than 20% of these fractures meet operative indications. Unfortunately, one of the major complications of these fractures is the development of avascular necrosis (AVN), or death of the bone as a result of the loss of blood supply to it. Currently, the ability to predict AVN is limited. The purpose of this study is to determine if computed tomography imaging can identify a quantifiable predictor of AVN following this type of humeral fracture.

DETAILED DESCRIPTION:
Current surgical treatment of humeral head fracture does not follow a universally accepted treatment algorithm. Treatment guidelines are lacking sufficient prospective controlled evidence to support any one option as doctrine. However, the generally accepted dogma regarding the surgical treatment of fractures considered high-risk for Avascular Necrosis (AVN), and also symptomatic avascular necrosis of the humeral head, is shoulder replacement (arthroplasty). This is a difficult scenario for younger patients where humeral head preservation is the priority, because of a expected lifespan that will require one, if not multiple, arthroplasty revisions. There is data suggesting no difference in functional outcome for complx humeral head fractures treated with open reduction and internal fixation (ORIF), that late progress to AVN, and patients who undergo hemi-arthroplasty, because of risk of AVN. However, failure of surgery related to AVN remains a challenging problem often leading to secondary surgery, which is not without negative outcomes. This study is aimed at trying to come up with a predictor that can be applied to patients prior to initial humeral head fracture treatment.

The specific aims of the study to help determine this predictor are:

1. In patients who have humeral head fracture, evaluate the difference in fracture fragment enhancement in multi-part fractures, by comparing the fracture fragment attenuation on iodine map overlay to the non-traumatized, contralateral humeral head using Dual Energy Computed Tomography (DECT).
2. In patients undergoing ORIF or joint replacement for humeral head fracture without known risk factors for AVN, identify the relationship between the attenuation due to iodine in the fractured humeral head, as measured preoperatively by DECT, with the presence of pulsatile blood flow in the humeral head intra-operatively, as measured with laser doppler.
3. In patients undergoing joint replacement for humeral head fracture without other known risk factors for AVN, identify the relationship between the attenuation due to iodine in the fractured humeral head, as measured preoperatively by DECT, with the presence of AVN in humeral head pathology specimen.
4. In patients who underwent ORIF for humeral head fracture without other known risk factors for AVN, identify the relationship between the attenuation due to iodine within the fractured humeral head, as measured preoperatively by DECT, with the incidence of radiographically apparent AVN after 2 years of clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multi-part fracture of proximal humerus.

Exclusion Criteria:

* Patients with a humeral head prosthesis, hardware or avascular necrosis in the ipsilateral shoulder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting adult patients with proximal humerus fractures.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Evidence of avascular necrosis post humeral head fracture. | Within 2 years of fracture correction or surgery.
  All patients who have humeral head fractures will have a dual energy CT examination performed with intravenous contrast to evaluate the fracture pattern to determine if the patient is a surgical candidate. The amount of contrast within the fractured humeral head will be measured on this CT scan as a surrogate for blood flow. After conservative (no surgery) or surgical (open reduction internal fixation) treatment, the patient will be followed in the orthopedics clinic for two years. During each twice yearly visit, shoulder radiographs will be obtained. Standardized criteria for radiograph assessment to determine AVN will be used: mixed lucent and sclerotic appearance of the humeral head, subchondral collapse as indicated by a "crescent sign" and/or loss of humeral head sphericity. AVN will be described as present or absent based on the radiographic findings. The incidence of AVN will be correlated with the amount of contrast within the humeral head as measured by dual energy CT.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hoover, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Hoover KB, Starks AO, Robila V, Riddle DL. Quantitative contrast enhanced dual energy CT to predict avascular necrosis: a feasibility study of proximal humerus fractures. BMC Med Imaging. 2021 Dec 11;21(1):191. doi: 10.1186/s12880-021-00717-x. PMID 34895190